CLINICAL TRIAL: NCT04232293
Title: Screening of Liver Fibrosis Using Blood Tests in Patients With Type 2 Diabetes Mellitus
Acronym: L-FibroT2DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC19_0425
Record Dates: First submitted 2020-01-06; First posted 2020-01-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Diabetes Mellitus, Type 2; NAFLD; NASH
Keywords: NASH; NAFLD; Fibrosis; Cirrhosis; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease; Fibrosis | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood tests (Experimental): Two diagnostic tests (eLift and FibroMeter) will be performed to evaluate liver fibrosis
  Interventions: Diagnostic Test: Blood tests

INTERVENTIONS:
Diagnostic Test: Blood tests — eLift and FibroMeter

SUMMARY:
Non-Alcoholic Fatty Liver Disease (NAFLD) and Non-Alcoholic SteatoHepatitis (NASH), are a frequent complication of type 2 diabetes and obesity. This disease has been linked with an increased morbidity and mortality, in particular cardiovascular disease and hepatic complications (cirrhosis and hepatocellular carcinoma). NAFLD is covered different liver damage in ascending order: steatosis, Non-Alcoholic SteatoHepatitis (NASH), fibrosis, and finally cirrhosis. Mostly, fibrosis has a determining role in the patient's status health. The fibrosis prevalence rate may reach up to 15 % of people with type 2 diabetes. The purpose of the study is to screen hepatic fibrosis for patient with type 2 diabetes.

To be sure of the status of the disease, the gold standard procedure remains liver biopsy. However, it's an invasive procedure and it's a challenge to perform this kind of medical procedure to every patient with NAFLD. Some alternative procedure exists, called FibroScan that gives some indication of liver fibrosis status. Unfortunately, every diabetologist hasn't this equipment in his medical office. The investigators propose to evaluate two non-invasive biological fibrosis tests, called eLIFT and FibroMeter. The results of these two diagnostic tests will be compared to FibroScan and to liver biopsy results.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years old,
* Type 2 diabetes mellitus for more than 6 months,
* BMI > 25 kg/m2,
* Waist circumference > 94 cm (male) or 80 cm (female).
* Patient benefiting from a social security system.

Exclusion Criteria:

* Medical follow up for liver disease,
* Decompensated cirrhosis,
* Health status that does not allow the participation of the patient,
* Hospitalisation for acute complication: sepsis, infection, foot's ulcer, acute coronary syndrome,…
* HbA1c > 11,0 %,
* Pregnancy.
* Patient under guardianship or curatorship or protection of justice
* Involvement refusal.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 722 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-06-27 (Actual)

PRIMARY OUTCOMES:
eLift and FibroMeter sensitivity for the diagnosis of advanced hepatic fibrosis | Day 0
  sensitivity calculated as follows: (number of patients with advanced hepatic fibrosis and a positive test) / (number of patients with advanced hepatic fibrosis)

SECONDARY OUTCOMES:
number of advanced hepatic fibrosis diagnosed according to the FibroScan composite criterion and then liver biopsy | 3 months
Controlled Attenuation Parameter (CAP) measurement by FibroScan | 3 months
Patient rate with eLIFT ≥8 versus FibroMeter ≥0.22. | Day 0
Liver hardness (kPa) measured by FibroScan | 3 months
Complication of diabetes | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand CARIOU, Pr, Principal Investigator — Nantes Hospital University
Locations (2):
- France (2):
  - CHU d'Angers, Angers
  - CHU de Nantes, Nantes

IPD SHARING:
Plan to Share IPD: No